CLINICAL TRIAL: NCT01265459
Title: Double-Blind, Randomized Study of Three Different Volumes of Durolane in Subjects With Osteoarthritis of the Knee
Brief Title: Different Volumes of Durolane in Knee OA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35GA1001
Record Dates: First submitted 2010-12-17; First posted 2010-12-23 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2014-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Durolane 3ml (Experimental): Durolane 3 ml is an Intraarticular hyaluronic acid
  Interventions: Device: Durolane 3 ml, Durolane 4,5 ml, Durolane 6 ml
- Durolane 4.5 (Experimental): Durolane 4.5 is an Intraarticular hyaluronic acid
  Interventions: Device: Durolane 3 ml, Durolane 4,5 ml, Durolane 6 ml
- Durolane 6 ml (Experimental): Durolane 6 ml is an Intraarticular hyaluronic acid
  Interventions: Device: Durolane 3 ml, Durolane 4,5 ml, Durolane 6 ml

INTERVENTIONS:
Device: Durolane 3 ml, Durolane 4,5 ml, Durolane 6 ml — Durolane is an intraarticular hyaluronic acid preparation

SUMMARY:
The purpose of the study is to assess the safety and efficacy profiles of new single-injection volumes of Durolane in patients with knee OA.

DETAILED DESCRIPTION:
To assess the safety and efficacy profiles of different volumes of Durolane in patients with knee OA and compare with the current standard single-injection of the product. The study aims to investigate whether different volumes of Durolane compared to the standard injection volume will improve the benefit/risk profile.

ELIGIBILITY:
Inclusion Criteria:

* Subject (female or male)
* 40-85 years of age
* Unilateral knee pain fulfilling American College of Rheumatology (ACR) criteria for diagnosis of osteoarthritis(OA)
* Radiographic evidence of OA in the study knee
* WOMAC pain score of 7-17 in the study knee
* WOMAC pain score of 2-3 in the study knee (WOMAC Likert 3.1 A1)
* Subject normally active
* Subject has attempted but not responded adequately to previous non-pharmacological therapy(ies)and to simple analgetics
* Subject cooperative and able to communicate effectively with the investigators
* Body mass index ≤ 35 kg/m2;
* Signed informed consent obtained

Exclusion Criteria:

* Knee effusion
* Contralateral knee OA
* Clinically significant joint pain from joints other than the knee
* Previous intra-articular steroid injection into the study knee within the last 6 months
* Previous intra-articular Hyaluronic Acid (HA) injection into the study knee within the last 9 months
* Previous allergic type reaction to a HA product
* Treatment with analgesics other than paracetamol (acetaminophen) (including topical agents for the knee) within 5 half lives of the drug prior to the baseline visit
* Use of analgesics 48 hours preceding the baseline visit
* Use of systemic glucocorticosteroids (excluding inhaled steroids) within the last 3 months
* Treatment with glucosamine/chondroitin sulfate initiated within the past 3 months
* Change in physical therapy for the knee within the last three months
* Arthroscopy or other surgical procedure in the study knee within the past 12 months
* Serious injuries to the study knee in the past
* Any planned arthroscopy or other surgical procedure during the study period
* Previous history or presence of active septic arthritis
* Active skin disease or infection in the area of the injection site
* Systemic active inflammatory condition or infection
* Bleeding diathesis or use of anticoagulants
* History of drug or alcohol abuse within 6 months
* Any medical condition that in the opinion of the investigator makes the subject unsuitable for inclusion
* Pregnant or breastfeeding woman or woman of childbearing potential not practicing adequate contraception
* Involvement in other clinical trials

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per-Erik Melberg, MD, Principal Investigator — Kristinelundskliniken, Kristinelundsgatan 13, 411 37 Göteborg
Locations (3):
- Sweden (3):
  - Torsten Adalberth, Malmo
  - Christian Akermark, Stockholm
  - Johan Isacson, Upplands Vasby

RESULTS

PARTICIPANT FLOW:
Groups:
- Durolane 3 mL: Single injection of 3 ml Durolane (Durolane is an intraarticular hyaluronic acid preparation)
- Durolane 4.5 mL: Single injection of 4.5 ml Durolane (Durolane is an intraarticular hyaluronic acid preparation)
- Durolane 6 mL: Single injection of 6 ml Durolane (Durolane is an intraarticular hyaluronic acid preparation)
Period: Overall Study
Arm/Group | Durolane 3 mL | Durolane 4.5 mL | Durolane 6 mL
Started | 23 | 23 | 22
Completed | 23 | 23 | 20
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Durolane 3 mL | Durolane 4.5 mL | Durolane 6 mL | Total
Number analyzed (Participants) | 23 | 23 | 22 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 22 | 68
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.8) | 64.1 (8.0) | 62.8 (7.3) | 63.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 10 | 32
  Male | 12 | 12 | 12 | 36
Region of Enrollment [Number; unit: participants]
  Sweden | 23 | 23 | 22 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain Over 26 Weeks (Change From Baseline)
Description: The study aims to compare the change of pain for different volumes of study product over 26 weeks using WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) pain score that consists of 5 questions.
  It is a 5-graded Likert scale: None, Mild, Moderate, Severe or Extreme relating to how much pain the subject has experienced during the last 48 hours. The score of each dimension is calculated by simply adding the score (from 0 to 4) for each question.
Time Frame: 26 weeks after treatment compared to baseline
Population: The primary population for all efficacy evaluations was the ITT population (all subjects randomized and treated with study product).
  No imputation of missing data was done. Analyses presented were based on observed cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Durolane 3 mL; Durolane 4.5 mL; Durolane 6 mL: WOMAC pain score at 26 weeks (change from baseline). Single intra-articular injection of Durolane (20mg/ml).
Arm/Group | Durolane 3 mL | Durolane 4.5 mL | Durolane 6 mL
Number analyzed (Participants) | 23 | 23 | 20
units on a scale | -4.13 (4.39) | -4.00 (3.74) | -4.90 (5.06)

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability From Baseline to 26 Weeks After Treatment.
Description: Safety and tolerability will be assessed at each clinic visit (Baseline, 2, 6, 12, 18 and 26 weeks). Standard questions was used, "Since your last clinical visit have you had any health problems?".
Time Frame: From baseline to 26 weeks after treatment
Measure: Number; unit: participants
Arm/Group | Durolane 3 mL | Durolane 4.5 mL | Durolane 6 mL
Number analyzed (Participants) | 23 | 23 | 20
participants | 8 | 12 | 14

3. Secondary Outcome: WOMAC Stiffness Score (Change From Baseline)
Description: The study aims to compare the change of stiffness for different volumes of study product over 26 weeks using WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) stiffness score that consists of 2 questions.
  It is a 5-graded Likert scale: None, Mild, Moderate, Severe or Extreme relating to how much stiffness the subject has experienced in the last 48 hours. The score of each dimension is calculated by simply adding the score (from 0 to 4) for each question.
Time Frame: 26 weeks after treatment compared to baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Durolane 3 mL; Durolane 4.5 mL; Durolane 6 mL: WOMAC stiffness score at 26 weeks (change from baseline). Single injection of Durolane (20 mg/ml).
Arm/Group | Durolane 3 mL | Durolane 4.5 mL | Durolane 6 mL
Number analyzed (Participants) | 23 | 23 | 20
units on a scale | -1.30 (2.27) | -1.39 (1.85) | -1.15 (1.90)

4. Secondary Outcome: WOMAC Physical Function Score (Change From Baseline)
Description: The study aims to compare the physical function for different volumes of study product over 26 weeks using WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) physical function score that consists of 17 questions.
  It is a 5-graded Likert scale: None, Mild, Moderate, Severe or Extreme relating to performing daily physical activities the subject has experienced in the last 48 hours. The score of each dimension is calculated by simply adding the score (from 0 to 4) for each question.
Time Frame: 26 weeks after treatment compared to baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Durolane 3 mL; Durolane 4.5 mL; Durolane 6 mL: WOMAC physical function score at 26 weeks (change from baseline). Single injection of Durolane (20 mg/ml).
Arm/Group | Durolane 3 mL | Durolane 4.5 mL | Durolane 6 mL
Number analyzed (Participants) | 23 | 23 | 20
units on a scale | -11.14 (13.98) | -13.13 (11.93) | -12.32 (14.86)

5. Secondary Outcome: Subject´s Global Assessment of the Status of the Study Knee (Change From Baseline)
Description: The subject will assess his/her global status how the study knee affects them by using a 11-point numerical rating scale, Subject global assessment scale, from "very poor=0" to "excellent=10".
Time Frame: 26 weeks after treatment compared to baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Durolane 3 mL; Durolane 4.5 mL; Durolane 6 mL: Subject´s global assessment of the status of the study knee at 26 weeks (change from baseline).
  Single injection of Durolane (20 mg/ml).
Arm/Group | Durolane 3 mL | Durolane 4.5 mL | Durolane 6 mL
Number analyzed (Participants) | 23 | 23 | 20
units on a scale | 1.43 (2.64) | 1.39 (2.44) | 1.70 (3.69)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected during 26 weeks.
Arm/Group | Durolane 3 mL | Durolane 4.5 mL | Durolane 6 mL
Serious Adverse Events (participants affected / at risk) | 0/23 | 2/23 | 1/22
Other Adverse Events (participants affected / at risk) | 8/23 | 12/23 | 14/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durolane 3 mL (N=23) | Durolane 4.5 mL (N=23) | Durolane 6 mL (N=22)
Pulmonary thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Headache and high fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal prolaps (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durolane 3 mL (N=23) | Durolane 4.5 mL (N=23) | Durolane 6 mL (N=22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (8) | 9 (9) — The related arthralgia events had a rapid onset and usually started within 1 day after injection of the study product and the duration was in general short.
Headache (Nervous system disorders) | 0 (0) | 4 (7) | 7 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less